CLINICAL TRIAL: NCT02558218
Title: Postoperative Discomfort and Ocular Redness Following Phacoemulsification and Intraocular Lens Implantation
Brief Title: Postoperative Discomfort and Ocular Redness Following Phacoemulsification Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FBCat
Record Dates: First submitted 2015-09-15; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — methylacetylene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane ultra group (Active Comparator): Participants in this group were administered systane ultra quid (Alcon, Fort Worth) for two months postoperatively), additionally to tobradex quid (Alcon, Fort Worth) for 20 days postoperatively.
  Interventions: Drug: Systane Ultra
- Control group (Active Comparator): Participants in this group were administered the standard postoperative medication [tobradex quid (Alcon, Fort Worth) for 20 days postoperatively.]
  Interventions: Drug: tobradex quid (Standard)

INTERVENTIONS:
Drug: Systane Ultra — Further to standard medication (tobradex quid for 20 days), participants were administered Systane Ultra quid for 2 months
  Other Names: Administration of Systane Ultra (Alcon)
  Arms: Systane ultra group
Drug: tobradex quid (Standard) — Standard medication (tobradex quid for 20 days)
  Other Names: Standard Medication
  Arms: Control group

SUMMARY:
Primary objective of the study is the assessment of the patients' discomfort and ocular redness following cataract extraction surgery by means of phacoemulsification and intraocular lens implantation.

DETAILED DESCRIPTION:
Participants will be recruited from the Cataract Service of the University Hospital of Alexandroupolis (UHA) in a consecutive-if-eligible basis. By means of a custom computer randomization program all participants will randomly populate either study group (who will receive Systane Ultra as additional postoperative treatment) and control group (who will receive standard postoperative treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of senile cataract with stage 2 or 3 nuclear opalescence according to the - Lens Opacities Classification System III (LOCS-3) grading scale

Exclusion Criteria:

1. Endothelial cell count less than 1900,
2. Glaucoma,
3. IOP-lowering medications,
4. Former incisional surgery,
5. Former diagnosis of corneal disease,
6. Diabetes or autoimmune diseases
7. Former diagnosis of dry eye disease

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Foreign body sensation | 1 month postoperatively
  Foreign body sensation will be assessed by a direct 5-scale, Likert type question that will be addressed to the participants at the 30th postoperative day

SECONDARY OUTCOMES:
Ocular Redness | 7 days postoperatively
  Ocular redness will be assessed by means of a validated photographic chart
Corneal Sensitivity | 1 month postoperatively
  Corneal Sensitivity will be assessed by Cochet-Bonnet esthesiometer at the 7th and 30th postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Eye Institute Of thrace, Alexandroupoli, Evros, Greece

REFERENCES:
- [Derived] Labiris G, Ntonti P, Sideroudi H, Kozobolis V. Impact of polyethylene glycol 400/propylene glycol/hydroxypropyl-guar and 0.1% sodium hyaluronate on postoperative discomfort following cataract extraction surgery: a comparative study. Eye Vis (Lond). 2017 May 10;4:13. doi: 10.1186/s40662-017-0079-5. eCollection 2017. PMID 28497070